CLINICAL TRIAL: NCT03233919
Title: Evaluation of Comprehensive Remote Ischemic Conditioning in ST-elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Brief Title: COmprehensive Remote Ischemic Conditioning in Myocardial Infarction
Acronym: CORIC-MI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, hongbing_yan, Co-Director, Center of cronary artery disease, Fuwai hospital, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-866
Record Dates: First submitted 2017-07-24; First posted 2017-07-31 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-03

CONDITIONS: Myocardial Infarction, Anterior Wall
Keywords: Remote Ischemic Conditioning
MeSH Terms: conditions — Anterior Wall Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CORIC (Experimental): Comprehensive remote ischaemic conditioning (CORIC) will be induced using an automated RIC device:
  Per-RIC consists of 5 cycles of 5-min inflation (200 mmHg) and 5-min deflation of cuff on a lower limb. The first inflation began immediately following randomization after admission. In case 5 cycles of RIC were not fully completed when the first balloon inflation or thrombus aspiration was ready to be performed, PCI was not to be delayed.
  Post-RIC consists of 5 cycles of 5-min inflation (200 mmHg) and 5-min deflation of cuff on a lower limb immediately after PPCI.
  Delayed-RIC consists of 5 cycles of 5-min inflation (200 mmHg) and 5-min deflation of cuff on a lower limb once daily on 2-28 days after MI.
  Interventions: Device: comprehensive remote ischaemic conditioning
- Non-CORIC (No Intervention): Controls did not undergo comprehensive remote ischaemic conditioning.

INTERVENTIONS:
Device: comprehensive remote ischaemic conditioning — comprehensive remote ischaemic conditioning will be induced using an automated RIC device: Per-RIC consists of 5 cycles of 5-min inflation (200 mmHg) and 5-min deflation of cuff on a lower limb. The first inflation began immediately following randomization after admission. In case 5 cycles of RIC were not fully completed when the first balloon inflation or thrombus aspiration was ready to be performed, PCI was not to be delayed.
  Post-RIC consists of 5 cycles of 5-min inflation (200 mmHg) and 5-min deflation of cuff on a lower limb immediately after PPCI.
  Delayed-RIC consists of 5 cycles of 5-min inflation (200 mmHg) and 5-min deflation of cuff on a lower limb once daily on 2-28 days after MI.
  Arms: CORIC

SUMMARY:
The primary objective of the CORIC-MI trial is to evaluate whether comprehensive (per, post plus delayed) remote ischemic conditioning (CORIC) as an adjunctive therapy in patients with ST-elevation myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention (PPCI) can improve left ventricular function and remodeling at 30 days assessed by cardiac magnetic resonance imaging (CMR) for a minimum follow-up period of 12 months.

DETAILED DESCRIPTION:
ST-segment elevation myocardial infarction (STEMI) is a leading cause of mortality and morbidity worldwide. Rapid admission and acute interventional treatment combined with modern antithrombotic pharmacologic therapy frequently establish complete reperfusion and acutely stabilize the patient, but the reperfusion itself adds further to the damage in the myocardium compromising the long-term outcome. At present, remote ischemic conditioning (RIC) is the most promising adjuvant therapy to reduce reperfusion injury in patients with STEMI. However, myocardial remodeling continues for several weeks after a myocardial infarction. Recent animal studies have shown that RIC may also help the heart muscle recover if applied every day during the month after a heart attack.

The CORIC-MI trial is a single-center, randomized, controlled, parallel group, and open-label trial, with blinded evaluation of the endpoints.The primary objective of the trial is to evaluate whether comprehensive (per, post plus delayed) remote ischemic conditioning (CORIC) as an adjunctive therapy in patients with STEMI undergoing primary percutaneous coronary intervention (PPCI) can improve left ventricular function and remodeling at 30 days assessed by cardiac magnetic resonance imaging (CMR) for a minimum follow-up period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Suspected anterior STEMI: new ST-elevation > 0.1 millivolt (mV) (≥ 0.2 mV in men or ≥ 0.15 mV in women in leads V2-V3) in > two contiguous leads in V1-V6; new or presumed new left bundle branch block;
* Symptom onset no more than 12 h before presentation and planned primary PCI;
* Age 18 to 75 years;
* Willingness and capability to provide informed consent.

Exclusion Criteria:

* Previous anterior myocardial infarction;
* Previous coronary artery bypass graft (CABG);
* Myocardial infarction or stroke within the previous 30 days;
* Treatment with thrombolysis within the previous 30 days;
* Cardiogenic shock;
* Thrombolysis in myocardial infarction (TIMI) flow grade 2 or 3 at coronary angiography;
* Coronary anatomy or mechanical complication of STEMI (ventricular septal rupture, free wall rupture, acute severe mitral regurgitation) warranting emergent surgery;
* Inability to obtain TIMI flow grade ≥ 2;
* Conditions precluding use of RIC (paresis of lower limb, known severe peripheral artery disease or evidence of lower limb ischemia, and etc.);
* Life expectancy of less than 12 months due to non-cardiac disease such as known malignancy or other comorbid conditions;
* Contraindications to CMR;
* Treated with therapeutic hypothermia before admission;
* Pregnancy and lactating women;
* Participation in another interventional trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-01-30 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
left ventricular ejection fraction (LVEF) assessed by CMR | at 30 days after MI
  LVEF assessed by CMR at 30 days

SECONDARY OUTCOMES:
Infarct size assessed by CMR. | at 30 days after MI
  Infarct size assessed by CMR delayed enhancement volume at 30 days.
LVEDVi and LVESVi assessed by CMR. | at 30 days after MI
  LVEDVi and LVESVi assessed by cMRI at 30 days
LVEF assessed by echocardiography. | at 30 days, 180 days and 365 days after MI
  LVEF assessed by echocardiography at 30 days, 180 days and 365 days.
LVEDVi assessed by echocardiography. | at 30 days, 180 days and 365 days after MI.
  LVEDVi assessed by echocardiography at 30 days, 180 days and 365 days.
The change in LVEDVi assessed by echocardiography. | at 30 days, 180 days and 365 days after MI.
  The change in LVEDVi assessed by echocardiography from baseline to 30 days, 180 days or 365 days.
MACE including death, re-infarction, rehospitalization for heart failure, and ischemic stroke | at 30 days, 180 days and 365 days after MI.
  MACE including death, re-infarction, rehospitalization for heart failure, and ischemic stroke at 30 days, 180 days and 365 days.
Mean blood N terminal (NT)-PROBNP levels | at 30 days, 180 days and 365 days
  Mean blood NT-PROBNP levels at 30 days, 180 days and 365 days.
TIMI flow and frame count | at the last angiogram during PPCI
  TIMI flow and frame count are evaluated at the last angiogram during PPCI.
ST-segment resolution | on 90 min ECG after reperfusion
  ST-segment resolution on 90 min ECG after reperfusion
the 6-min walk test distance | at 30 days and 180 days after MI
  the 6-min walk test distance at 30 days and 180 days after MI.
Mean Self-rating Anxiety Scale (SAS) score | at 30 days and 180 days after MI
  Mean SAS score at 30 days and 180 days after MI.
Mean Self-rating Depression Scale (SDS) score | at 30 days and 180 days after MI.
  Mean SDS score at 30 days and 180 days after MI.
Mean score of health-related quality of life by using Short-Form 36 Health Survey (SF-36). | at 30 days and 180 days after MI.
  The mean score of health-related quality of life by using SF-36 at 30 days and 180 days after MI.

OTHER OUTCOMES:
Contrast-induced nephropathy | at 72 hour and 30 days post-PPCI
  Contrast-induced nephropathy at 72 hour and 30 days post-PPCI
Platelet reactivity | at baseline, 6 hours post-loading dose of antiplatelet, 7 days, 30 days and 180 days after MI.
  Platelet reactivity assessed by VerifyNow P2Y12 assay at baseline, 6 hours post-loading dose of antiplatelet, 7 days, 30 days and 180 days after MI.

CONTACTS AND LOCATIONS:
Overall Officials: hongbing Yan, MD, Principal Investigator — National Center for Cardiovascular Diseases; Chinese Academy of Medical Sciences, Fuwai Hospital, Principal Investigator — National Center for Cardiovascular Diseases
Locations (1):
- Chinese Academy of Medical Sciences, Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No